CLINICAL TRIAL: NCT02151617
Title: A Phase 1 Double Blind (3rd Party Open) Randomized, Placebo Controlled, Dose Escalation Study To Investigate The Safety,Tolerability, Pharmacokinetics And Pharmacodynamics Of Repeat Doses Of Pf-06743649 With Or Without Food In Healthy Adult Subjects
Brief Title: A Study In Healthy People To Evaluate Safety, Toleration, Pharmacokinetics And Pharmacodynamics Of Multiple Oral Doses Of PF-06743649
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7911001
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
Keywords: Multiple dose; safety; tolerability; PK

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1-PF-06743649 or placebo (Experimental): Subjects will be randomized to receive PF-06743649 or placebo as 2 single doses in periods 1 and 2 either in the fed or fasted state followed by once daily dosing for 14 days in period 3
  Interventions: Drug: PF-06743649; Drug: Placebo
- Cohort 2-PF-06743649 or placebo (Experimental)
  Interventions: Drug: PF-06743649; Drug: Placebo
- Cohort 3-PF-06743649 or placebo (Experimental)
  Interventions: Drug: PF-06743649; Drug: Placebo
- Cohort 4-PF-06743649 or placebo (Experimental)
  Interventions: Drug: PF-06743649; Drug: Placebo
- Cohort 5-PF-06743649 or placebo (Experimental)
  Interventions: Drug: PF-06743649; Drug: Placebo

INTERVENTIONS:
Drug: PF-06743649 — 40 mg tablet one time once with a meal and once without a meal, followed by once daily dosing for 14 days
  Arms: Cohort 1-PF-06743649 or placebo
Drug: Placebo — Placebo tablet one time once with a meal and once without a meal, followed by once daily dosing for 14 days
  Arms: Cohort 1-PF-06743649 or placebo
Drug: PF-06743649 — To be decided dose, tablet once daily dosing for 14 days
  Arms: Cohort 2-PF-06743649 or placebo
Drug: Placebo — Placebo tablet once daily dosing for 14 days
  Arms: Cohort 2-PF-06743649 or placebo
Drug: PF-06743649 — To be decided dose, tablet, one time once with a meal and once without a meal, followed by once daily dosing for 14 days
  Arms: Cohort 3-PF-06743649 or placebo
Drug: Placebo — Placebo tablet one time once with a meal and once without a meal, followed by once daily dosing for 14 days
  Arms: Cohort 3-PF-06743649 or placebo
Drug: PF-06743649 — To be decided dose, tablet, one time without a meal, followed by once daily dosing for 14 days
  Arms: Cohort 4-PF-06743649 or placebo
Drug: Placebo — Placebo tablet one time once without a meal, followed by once daily dosing for 14 days
  Arms: Cohort 4-PF-06743649 or placebo
Drug: PF-06743649 — Tablet, to be decided dose, once daily, 14 days
  Arms: Cohort 5-PF-06743649 or placebo
Drug: Placebo — Tablet, once daily, 14 days
  Arms: Cohort 5-PF-06743649 or placebo

SUMMARY:
The purpose of this study in healthy people is to evaluate safety, toleration and time course of plasma concentration of multiple oral doses of PF-06743649. The pharmacodynamic activity of PF-06743649 will also be assessed. The effect of food on PK of PF-06743649 will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* Evidence of gout/hyperuricemia, measured sUA >8 mg/dL at screening.
* Experienced an episode of nephrolithiasis or ureterolithiasis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | up to 14 days
Area Under the Curve from Time Zero to end of dosing interval (AUCtau) | up to 14 days
Time to Reach Maximum Observed Plasma Concentration (Tmax) | up to 14 days
Plasma Decay Half-Life (t1/2) | up to 14 days
Amount of drug recovered unchanged in urine during the dosing interval (Aetau) | up to 14 days
Percent of dose recovered unchanged in urine during the dosing interval(Aetau%) | up to 14 days
Renal clearance (CLr) | up to 14 days

SECONDARY OUTCOMES:
Change from baseline in serum uric acid level | up to 14 days
Change from baseline in serum levels of xanthine and hypoxanthine | up to 14 days
Urinary uric acid levels | up to 14 days
Urinary xanthine levels | up to 14 days
Urinary hypoxanthine levels | up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7911001&StudyName=A%20Study%20In%20Healthy%20People%20To%20Evaluate%20Safety%2C%20Toleration%2C%20Pharmacokinetics%20And%20Pharmacodynamics%20Of%20Multiple%20Oral%20Doses%20Of%20PF-06743649